CLINICAL TRIAL: NCT02462551
Title: Investigating the Effects of Focal Electrically Administered Seizure Therapy (FEAST) for the Treatment of Depression
Brief Title: Focal Electrically Administered Seizure Therapy for the Treatment of Depression
Acronym: FEAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziad Nahas (Other)
Collaborators: Columbia University (Other); MECTA corporation (Unknown); Medical University of South Carolina (Other)
Responsible Party: Sponsor-Investigator, Ziad Nahas, Professor and Chair of the Department of Psychiatry, American University of Beirut Medical Center
Organization: American University of Beirut Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21024/ PSY.ZN.03
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Treatment-Resistant Depression
Keywords: Depression; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FEAST (Experimental): Patients with treatment-resistant depression will undergo 3 sessions of focal electrically administered seizure therapy for two to six weeks. The complete parameter range of the stimulus delivered (Freq: 20-120 Hz; PW: 0.2-2 ms; Duration: 0.1 to 8 s; Current: 0.5-0.8A; charge: 1-576 mC) is determined by an initial titration session and the PI (as an expert in neuromodulation treatments).
  Interventions: Device: Focal Electrically Administered Seizure Therapy

INTERVENTIONS:
Device: Focal Electrically Administered Seizure Therapy — A focal administration of the right unilateral configuration of electro-convulsive therapy for the treatment of recurrent and treatment-resistant depression.
  Other Names: FEAST

SUMMARY:
The purpose of this study is to determine the efficacy and any possible side effects of focal electrically administered seizure therapy (FEAST) as a treatment intervention for patients with recurrent and treatment resistant depression.

DETAILED DESCRIPTION:
Recurrent and treatment resistant depression (TRD) has high morbidity and escalating costs for the healthcare system and society at large. Electroconvulsive therapy (ECT) remains the most effective acute antidepressant treatment for TRD, but with significant risks of cognitive impairment. The efficacy and side effects of conventional ECT are contingent on the anatomic positioning of electrodes and stimulus dosage. A technique that could spatially target the prefrontal cortex may preserve the efficacy of ECT while simultaneously reducing cognitive side effects.

The investigators have recently demonstrated that focal electrically-administered seizure therapy [FEAST], which markedly improves the spatial targeting of the electrical current, is feasible in adult TRD individuals. FEAST can initiate seizures focally and specifically in the prefrontal cortex prior to secondary seizure generalization. Preliminary results in depressed humans at Columbia University and later at the Medical University of South Carolina (MUSC) generated by the PI (Nahas) show that these focal seizures produce clinically meaningful antidepressant responses. Additional work is needed to refine the technique and compare it to conventional approaches.

In this study, the investigators will further develop FEAST to achieve clinically meaningful remission rates (at least 50% of subjects). 30 TRD patients (or 20 with a complete record) will undergo an open-label course of FEAST for an adaptive number of total sessions designed to maximize efficacy of the technique. The investigators will use a dosing paradigm using a current level of 800 mA, finalize the electrode sizes, and test, at one treatment session, the effects of reversing the directionality of current flow on site of seizure induction. Patients will also undergo electroencephalography (EEG) assessments to characterize the induced seizures' spatial and temporal distributions. The investigators will obtain time to orientation recovery as a marker of potential longer-term cognitive side effects.

This technique could fundamentally change and improve the most effective antidepressant treatment, while simultaneously minimizing or eliminating the major side-effects that prohibit larger adoption of ECT.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years (inclusive)
* Diagnosis of major depressive disorder (unipolar or bipolar) [SCID to derive RDC; DSM-IV]
* Pretreatment HRSD score ≥ 18 [Hamilton Rating Scale for Depression (24-item)]
* ECT indicated [Physician evaluation]
* Willing and capable of providing informed consent [Physician evaluation]

Exclusion Criteria:

* History of schizophrenia, schizoaffective disorder, other functional psychosis, or rapid cycling bipolar disorder [SADS to derive RDC; rapid cycling defined as ≥ four episodes in past year]
* History of neurological illness or insult other than conditions associated with psychotropic exposure (e.g., tardive dyskinesia) [Physician evaluation; medical history]
* Alcohol or substance abuse or dependence in the past year (RDC) [Physician evaluation]
* Secondary diagnosis of a delirium, dementia, or amnestic disorder (DSM-IV), pregnancy, or epilepsy [Physician evaluation]
* Requires especially rapid antidepressant response due to suicidality, psychosis, inanition, psychosocial obligations, etc. [Physician evaluation]
* Unable to tolerate psychotropic washout and no psychotropic medication during the ECT trial, other than lorazepam (up to 3 mg/d PRN) [Treatment history and physician evaluation]
* ECT in the past six months [Physician evaluation; medical history]
* Has a cardiovascular and/or pulmonary condition [Physician evaluation]

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Spatial and temporal distribution and power of induced seizure on EEG recordings | 15 min before to 5 min after stimulus delivery for the first 3 sessions in a maximum period of two weeks
  EEG recordings will be analyzed to assess the dynamics and characteristics of induced seizure activity; including spatial and temporal distribution, power, and current density in different cortical areas

SECONDARY OUTCOMES:
Change in Depression Scores | Baseline and 4-6 weeks
  24-item Hamilton Depression Rating Scale
Time for Reorientation | 30 minutes
  Five questions are asked after waking up from anesthesia to assess short and long-term memory.

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Nahas, MD, MSCR, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Beyrouth, Lebanon

REFERENCES:
- [Background] Spellman T, Peterchev AV, Lisanby SH. Focal electrically administered seizure therapy: a novel form of ECT illustrates the roles of current directionality, polarity, and electrode configuration in seizure induction. Neuropsychopharmacology. 2009 Jul;34(8):2002-10. doi: 10.1038/npp.2009.12. Epub 2009 Feb 18. PMID 19225453
- [Background] Lisanby SH, Maddox JH, Prudic J, Devanand DP, Sackeim HA. The effects of electroconvulsive therapy on memory of autobiographical and public events. Arch Gen Psychiatry. 2000 Jun;57(6):581-90. doi: 10.1001/archpsyc.57.6.581. PMID 10839336
- [Background] Sackeim HA, Luber B, Moeller JR, Prudic J, Devanand DP, Nobler MS. Electrophysiological correlates of the adverse cognitive effects of electroconvulsive therapy. J ECT. 2000 Jun;16(2):110-20. doi: 10.1097/00124509-200006000-00003. PMID 10868321
- [Background] George MS, Nahas Z, Li X, Kozel FA, Anderson B, Yamanaka K, Chae JH, Foust MJ. Novel treatments of mood disorders based on brain circuitry (ECT, MST, TMS, VNS, DBS). Semin Clin Neuropsychiatry. 2002 Oct;7(4):293-304. doi: 10.1053/scnp.2002.35229. PMID 12382211
- [Background] Nahas Z, Short B, Burns C, Archer M, Schmidt M, Prudic J, Nobler MS, Devanand DP, Fitzsimons L, Lisanby SH, Payne N, Perera T, George MS, Sackeim HA. A feasibility study of a new method for electrically producing seizures in man: focal electrically administered seizure therapy [FEAST]. Brain Stimul. 2013 May;6(3):403-8. doi: 10.1016/j.brs.2013.03.004. Epub 2013 Mar 16. PMID 23518262
- [Background] Chahine G, Short B, Spicer K, Schmidt M, Burns C, Atoui M, George MS, Sackeim HA, Nahas Z. Regional cerebral blood flow changes associated with focal electrically administered seizure therapy (FEAST). Brain Stimul. 2014 May-Jun;7(3):483-5. doi: 10.1016/j.brs.2014.02.011. Epub 2014 Feb 22. PMID 24795198
- [Background] Nobler MS, Luber B, Moeller JR, Katzman GP, Prudic J, Devanand DP, Dichter GS, Sackeim HA. Quantitative EEG during seizures induced by electroconvulsive therapy: relations to treatment modality and clinical features. I. Global analyses. J ECT. 2000 Sep;16(3):211-28. doi: 10.1097/00124509-200009000-00002. PMID 11005043
- [Background] Luber B, Nobler MS, Moeller JR, Katzman GP, Prudic J, Devanand DP, Dichter GS, Sackeim HA. Quantitative EEG during seizures induced by electroconvulsive therapy: relations to treatment modality and clinical features. II. Topographic analyses. J ECT. 2000 Sep;16(3):229-43. doi: 10.1097/00124509-200009000-00003. PMID 11005044
- [Background] Kayser S, Bewernick BH, Grubert C, Hadrysiewicz BL, Axmacher N, Schlaepfer TE. Antidepressant effects, of magnetic seizure therapy and electroconvulsive therapy, in treatment-resistant depression. J Psychiatr Res. 2011 May;45(5):569-76. doi: 10.1016/j.jpsychires.2010.09.008. Epub 2010 Oct 16. PMID 20951997